CLINICAL TRIAL: NCT06466252
Title: Development and Psychometric Testing of a Questionnaire to Assess HPV Knowledge in Indonesia
Brief Title: Development and Psychometric Testing of HPV Knowledge Scale
Status: Completed | Type: Observational
Sponsor: Kaohsiung Medical University (Other)
Responsible Party: Principal Investigator, Yudisa Diaz Lutfi Sandi, Principal Investigator, Kaohsiung Medical University
Other Study IDs: 421/061/404.102.28/II/2023
Record Dates: First submitted 2024-06-11; First posted 2024-06-20 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Parents; Parent-Child Relations
Keywords: Human papillomavirus; parent; knowledge; Instrument development; psychometric test

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Psychometric Group — There are no interventions

SUMMARY:
The aim of this study is to develop and conduct psychometric testing of a new scale, the Human Papillomavirus Knowledge Scale (HPV-KS), particularly designed to assess HPV knowledge among parents of school-age children in Indonesia.

DETAILED DESCRIPTION:
research process after obtaining school principal. because the target population was parents who have daughters in elementary schools.

All participants (parents) were recruited from 5 elementary schools. According to a minimum sample size estimation for a psychometric study, it needs 10 times the total number of items (Boateng, 2018). the total participants, 52 items x 10= 520 participants were required.

The researchers got approval from schools to invite parents to attend the school of event invitations. Each participant came to the school where their child attended. Parents attended the regular meeting on the appointed day. at that time, researchers approached potential participants to explain to them the purpose of this study, participant rights, risks, and benefits. The researcher obtained participants' consent to participate in this research with a serial number.

During the process, researchers keep the participant anonymous. The questionnaires were distributed to the participants and took around 15-20 minutes to complete. All data was recapitulated and stored in Excel format. Data were kept by the researcher to maintain confidentiality. All data analyses were performed using SPSS software from IBM Corp.

Statistical analyses are below:

1. Descriptive analysis was used to identify population characteristics
2. Validity testing contains Exploratory and Confirmatory factor analyses were structure and construct.
3. Reliability testing was done using Cronbach alpha to determine the instrument's reliability.

ELIGIBILITY:
Inclusion Criteria:

* Participants have a child in elementary school
* Participants could speak Bahasa Indonesia fluently
* Participants live with their children in one house
* Participants are willing to participate in the study

Exclusion Criteria:

* parents had mental, visual, and hearing impairments or problems diagnosed by doctors
* their children' age are over 14 years old.

Min Age: 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All participants were parents who had children in elementary school. they come from several different educational variations, ethnicities, religions, places of residence, and economic levels. This research involved five elementary schools in rural areas. The population in rural was chosen to provide an overview of the understanding of rural communities regarding the feasibility of this new instrument.
Sampling Method: Non-Probability Sample
Enrollment: 673 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
Human papillomavirus knowledge scale | one time collected. participants took 15 minutes to complete all items in form.
  it consists of 3 subscales assessed awareness and understanding about human papillomavirus that encompass transmission, related to diseases, prevention, vaccine domestic policy context. it has a binary response format with a true /false response. the items contain favourable and unfavourable statement. A 1-point reflects that the answer is correct and 0-point is incorrect answer. The total scores indicated the knowledge level. The higher score means a better knowledge level

CONTACTS AND LOCATIONS:
Locations (1):
- Elementary school, Ngawi, East Java, Indonesia

REFERENCES:
- [Result] Hoppe-Seyler K, Bossler F, Braun JA, Herrmann AL, Hoppe-Seyler F. The HPV E6/E7 Oncogenes: Key Factors for Viral Carcinogenesis and Therapeutic Targets. Trends Microbiol. 2018 Feb;26(2):158-168. doi: 10.1016/j.tim.2017.07.007. Epub 2017 Aug 17. PMID 28823569
- [Result] Li Y, Xu C. Human Papillomavirus-Related Cancers. Adv Exp Med Biol. 2017;1018:23-34. doi: 10.1007/978-981-10-5765-6_3. PMID 29052130
- [Result] Songane M, Grossmann V. The patent buyout price for human papilloma virus (HPV) vaccine and the ratio of R&D costs to the patent value. PLoS One. 2021 Jan 11;16(1):e0244722. doi: 10.1371/journal.pone.0244722. eCollection 2021. PMID 33428667
- [Result] Meites E, Szilagyi PG, Chesson HW, Unger ER, Romero JR, Markowitz LE. Human Papillomavirus Vaccination for Adults: Updated Recommendations of the Advisory Committee on Immunization Practices. MMWR Morb Mortal Wkly Rep. 2019 Aug 16;68(32):698-702. doi: 10.15585/mmwr.mm6832a3. PMID 31415491
- [Result] Garg A, Wheldon CW, Galvin AM, Moore JD, Griner SB, Thompson EL. The Development and Psychometric Evaluation of the Mid-adult Human Papillomavirus Vaccine Knowledge Scale in the United States. Sex Transm Dis. 2022 Jun 1;49(6):423-428. doi: 10.1097/OLQ.0000000000001615. Epub 2022 Feb 8. PMID 35608097
- [Result] Harrison SE, Yelverton V, Wang Y, Ostermann J, Fish LJ, Williams CL, Vasudevan L, Walter EB. Examining Associations between Knowledge and Vaccine Uptake Using the Human Papillomavirus Knowledge Questionnaire (HPV-KQ). Am J Health Behav. 2021 Sep 30;45(5):810-827. doi: 10.5993/AJHB.45.5.2. PMID 34702429
- [Result] Waller J, Ostini R, Marlow LA, McCaffery K, Zimet G. Validation of a measure of knowledge about human papillomavirus (HPV) using item response theory and classical test theory. Prev Med. 2013 Jan;56(1):35-40. doi: 10.1016/j.ypmed.2012.10.028. Epub 2012 Nov 8. PMID 23142106
- [Result] Trevisol FS, Nunes RD, Parma GOC, Manoel AL, Zapelini CM, Trevisol DJ, Traebert J. Internal construct validity of the Brazilian version of a tool for assessing the population's knowledge of human papillomavirus. Rev Bras Epidemiol. 2020 Jun 5;23:e200054. doi: 10.1590/1980-549720200054. eCollection 2020. PMID 32520104
- [Result] Sethi S, Santiago PHR, Soares GH, Ju X, Antonsson A, Canfell K, Smith M, Garvey G, Hedges J, Jamieson L. Development and validation of an HPV infection knowledge assessment scale among Aboriginal and Torres Strait Islander Peoples. Vaccine X. 2023 May 24;14:100317. doi: 10.1016/j.jvacx.2023.100317. eCollection 2023 Aug. PMID 37288370
- [Result] Grace-Leitch L, Shneyderman Y. Using the Health Belief Model to Examine the Link between HPV Knowledge and Self-Efficacy for Preventive Behaviors of Male Students at a Two-Year College in New York City. Behav Med. 2016 Jul-Sep;42(3):205-10. doi: 10.1080/08964289.2015.1121131. PMID 27337625
- [Result] Guvenc G, Seven M, Akyuz A. Health Belief Model Scale for Human Papilloma Virus and its Vaccination: Adaptation and Psychometric Testing. J Pediatr Adolesc Gynecol. 2016 Jun;29(3):252-8. doi: 10.1016/j.jpag.2015.09.007. Epub 2015 Sep 26. PMID 26409648
- [Result] Krawczyk A, Perez S, King L, Vivion M, Dube E, Rosberger Z. Parents' decision-making about the human papillomavirus vaccine for their daughters: II. Qualitative results. Hum Vaccin Immunother. 2015;11(2):330-6. doi: 10.4161/21645515.2014.980708. PMID 25692507
- [Result] Sinshaw MT, Berhe S, Ayele SG. Knowledge and Attitude Towards Human Papillomavirus Vaccine and Associated Factors Among Mothers Who Have Eligible Daughters in Debre Markos Town, Northwest Ethiopia. Infect Drug Resist. 2022 Mar 3;15:781-793. doi: 10.2147/IDR.S352440. eCollection 2022. PMID 35264861
- [Result] Pelullo CP, Di Giuseppe G, Angelillo IF. Human papillomavirus infection: knowledge, attitudes, and behaviors among lesbian, gay men, and bisexual in Italy. PLoS One. 2012;7(8):e42856. doi: 10.1371/journal.pone.0042856. Epub 2012 Aug 8. PMID 22905178
- [Result] Ojeaga A, Alema-Mensah E, Rivers D, Azonobi I, Rivers B. Racial Disparities in HPV-related Knowledge, Attitudes, and Beliefs Among African American and White Women in the USA. J Cancer Educ. 2019 Feb;34(1):66-72. doi: 10.1007/s13187-017-1268-6. PMID 28808906
- [Result] Forster AS, McBride KA, Davies C, Stoney T, Marshall H, McGeechan K, Cooper SC, Skinner SR. Development and validation of measures to evaluate adolescents' knowledge about human papillomavirus (HPV), involvement in HPV vaccine decision-making, self-efficacy to receive the vaccine and fear and anxiety. Public Health. 2017 Jun;147:77-83. doi: 10.1016/j.puhe.2017.02.006. Epub 2017 Mar 18. PMID 28404501